CLINICAL TRIAL: NCT03270111
Title: High Energy Expenditure From Physical Activity During a Weight Loss Intervention for Breast Cancer Survivors and High Risk Women
Brief Title: High Physical Activity During a Weight Loss Intervention for Breast Cancer Survivors and High Risk Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00141301
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Female
Keywords: breast cancer survivor; weight loss program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A2: Breast Cancer Survivor (Experimental): Participants will include breast cancer survivors who take part in a weight loss intervention program. The intervention is the same for all participants.
  Interventions: Behavioral: Supervised Exercise; Behavioral: Home-based Exercise; Behavioral: Reduced Energy Diet; Behavioral: Group Phone Calls
- B: High Risk Women (Experimental): Participants will include women at high risk of breast cancer who take part in a weight loss intervention program. The intervention is the same for all participants.
  Interventions: Behavioral: Supervised Exercise; Behavioral: Home-based Exercise; Behavioral: Reduced Energy Diet; Behavioral: Group Phone Calls

INTERVENTIONS:
Behavioral: Supervised Exercise — Participants will take part in supervised exercise activities two times per week at a YMCA. Length of the activity will be increased during participation in study. Participants will start at 40 minutes per week and work their way up to 120 minutes per week.
Behavioral: Home-based Exercise — Aerobic exercise activities to be completed at home. Participants will be asked to start out doing 60 minutes at home and work up to 180 minutes of purposeful aerobic home exercise per week.
Behavioral: Reduced Energy Diet — Diet is a nutritionally balanced, reduced energy diet recommended by the Academy of Nutrition and Dietetics.
Behavioral: Group Phone Calls — Sessions are weekly months 1-3 and every other week months 4-6. The calls will discuss lifestyle changes specific to participants and cover the effects of diet, physical activity, and weight on breast cancer risk, as well as body image and emotional eating.

SUMMARY:
The purpose of this second pilot study is to extend the feasibility demonstrated in NCT02963740 that the intervention achieves high levels of moderate to vigorous physical activity (MVI PA) and modulates risk biomarkers for breast cancer and cardiovascular disease in older, obese sedentary breast cancer survivors who are undergoing moderate calorie restriction.

DETAILED DESCRIPTION:
All subjects participate in same intervention. Intervention consists of a 6-month structured weight loss program utilizing portion controlled meals and a prescribed level of graduated physical activity with an eventual goal of 200 minutes or more per week. The program will include twice weekly sessions with a trainer at a local YMCA, and weekly phone group sessions the first 3 months with transition to unsupervised exercise and less frequent group phone sessions the second 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer having completed any cytotoxic chemotherapy, radiation or surgery at least 3 months prior to study entry (Cohort A2) OR No prior diagnosis of breast cancer but at high risk for development of breast cancer and participating in HSC 4601 (Cohort B)
* Body Mass Index (BMI) >30 kg/m2. Women with a BMI > 45 kg/m2 must be age < 60 and ability to perform physical activity must be confirmed
* By self-assessment, currently performing 60 minutes or less of purposeful exercise per week but able to walk at least 30 minutes on a level surface
* Possession of smart phone capable of running MyFitnessPal and Garmin Connect apps and willing to have diet and exercise data accessed by study personnel
* Access to a personal computer
* Live in the greater Kansas City Metropolitan Area
* Willing and able to perform moderate intensity exercise at least 5 days per week for 6 months. This consists of a supervised exercise intervention at one of the 15 YMCAs affiliated with our program for 2 days per week. Must be willing to perform unsupervised home exercise for the entire 6 months.
* Willing to participate in a weekly behavioral modification group phone call for first 3 months and every 2 weeks for the second 3 months
* Willing to participate in a controlled dietary intervention with portion controlled meals and partial meal replacements plus 35 servings of fruits and vegetables/week for 6 months and track food intake and exercise
* Blood tests (Cohort A2) must have been performed after completion of any breast cancer surgery, radiation therapy, or cytotoxic chemotherapy, with reasonably normal liver and renal function as well as a hemoglobin of 10 or higher and/or performed within a year of study entry

Exclusion Criteria:

* Use of metformin, insulin, steroids or prescription weight loss or anti-psychotic drugs within the prior 3 weeks
* Individuals with prior gastric bypass surgery or procedure that would impair absorption of nutrients
* Need for chronic immunosuppressive drugs
* Participation within the past 6 months on a structured weight loss program such as Weight Watchers®
* Physical impairments (bad hip, knees, feet, peripheral neuropathy) that would prohibit performing moderate intensity exercise at least 5 days per week.
* Any other condition or intercurrent illness that in the opinion of the investigator makes the subject a poor candidate for participation in the trial such as recent cardiac event
* Currently receiving investigational agents in a clinical trial

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Adherence to supervised exercise sessions | Week 12
  Adherence is defined as the percent of monitored sessions at the YMCA attended by the participant.

SECONDARY OUTCOMES:
Percent participants meeting physical activity goal | Week 12
  Measured as percentage of participants meeting final physical activity goal between week 9 to week 12. Measurement based off activity tracker participants will wear.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fabian CJ, Klemp JR, Marchello NJ, Vidoni ED, Sullivan DK, Nydegger JL, Phillips TA, Kreutzjans AL, Hendry B, Befort CA, Nye L, Powers KR, Hursting SD, Giles ED, Hamilton-Reeves JM, Li B, Kimler BF. Rapid Escalation of High-Volume Exercise during Caloric Restriction; Change in Visceral Adipose Tissue and Adipocytokines in Obese Sedentary Breast Cancer Survivors. Cancers (Basel). 2021 Sep 28;13(19):4871. doi: 10.3390/cancers13194871. PMID 34638355